CLINICAL TRIAL: NCT01866150
Title: A Retrospective Chart Review on the Use of Biologics in Monotherapy for the Treatment of Rheumatoid Arthritis: A Comparison of the Effectiveness of Biologic Monotreatment and Biologic and Methotrexate (MTX) Combination Treatment
Brief Title: A Retrospective, Observational Chart Review of Biologics in Monotherapy Versus the Combination Biologic Plus Methotrexate in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28642
Record Dates: First submitted 2013-05-21; First posted 2013-05-31 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This cross-sectional, non-interventional, retrospective chart review will compare the efficacy and safety of biologic monotherapy and biologic and methotrexate combination therapy in patients with rheumatoid arthritis who have had an inadequate response to prior treatment with disease-modifying anti-rheumatic drugs including methotrexate. Data will be collected from patients who have been on first-line biologic treatment for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Diagnosis of rheumatoid arthritis by a rheumatologist
* Patients who have responded inadequately to methotrexate or disease-modifying anti-rheumatic drugs (DMARDs) and are being prescribed a biologic in monotherapy or in combination with methotrexate and other classical DMARDs as per NICE guidelines

Exclusion Criteria:

* Primary diagnosis of a condition other than rheumatoid arthritis
* Current treatment with a biologic in combination without methotrexate
* Prior treatment with an experimental agent for rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis with an inadequate response to at least 2 DMARD treatments, one of which includes methotrexate, who are being treated with first-line biologic therapy
Sampling Method: Probability Sample
Enrollment: 476 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- United Kingdom (14):
  - Cambridge
  - Chelmsford
  - Cosham
  - Derby
  - Dudley
  - Edinburgh
  - Harlow
  - London
  - Newcastle upon Tyne
  - Norwich
  - Portadown
  - Stoke-on-Trent
  - Truro
  - Wigan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Retrospective data was collected for 450 participants of whom 151 received biologic monotherapy, 289 received biologic combination therapy and 10 could not be categorized. Participant flow and baseline characteristics are presented for overall population and endpoints are presented for individual group.
Groups:
- Overall Population: Retrospective chart review of all participants with rheumatoid arthritis (RA) who were being treated with first-line biologic drug therapy (any) as monotherapy or biologic combination therapy according to National Institute for Health and Care Excellence (NICE) guidelines. Biologic combination therapy included biologic drug therapy (any) plus methotrexate (MTX) or biologic plus MTX plus any other and classical disease-modifying antirheumatic drugs (DMARDs).
Period: Overall Study
Arm/Group | Overall Population
Started | 450
Completed | 450
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants entered analysis set: All participants entered in this retrospective chart review were included.
Groups:
- Overall Population: Retrospective chart review of all participants with RA who were being treated with first-line biologic drug therapy (any) as monotherapy or biologic combination therapy according to NICE guidelines. Biologic combination therapy included biologic drug therapy (any) plus MTX or biologic plus MTX plus any other and classical DMARDs.
Arm/Group | Overall Population
Number analyzed (Participants) | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 331
  Male | 119

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Disease Activity Score Based on 28-joint Count (DAS-28) and Erythrocyte Sedimentation Rate (DAS28-ESR) Remission at 6 Months (DAS28<2.6)
Description: The DAS28 score is a measure of the participant's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], participant's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. DAS28 equals (=) (0.56 multiplied by [*] the square root [√] of TJC) plus (+) (0.28 * √ of SJC) + (0.70 * the natural logarithm [ln] ESR in millimeters per hour [mm/h]) + (0.014 * participant's global assessment of disease activity). DAS28 Remission is defined as a DAS28 score <2.6.
Time Frame: Month 6
Population: Ten participants from all participants entered analysis set who could not be categorized as under biologic monotherapy or biologic combination therapy were excluded from analysis. Number of participants analyzed=participants with available data for DAS28-ESR at Month 6.
Measure: Number; unit: percentage of participants
Groups:
- Biologic Monotherapy: Retrospective chart review of participants with RA who were being treated with first-line biologic drug therapy (any) as monotherapy according to NICE guidelines.
- Biologic Combination: Retrospective chart review of participants with RA who were being treated with first-line biologic drug therapy (any) plus MTX or biologic plus MTX plus any other classical DMARDs according to NICE guidelines.
Arm/Group | Biologic Monotherapy | Biologic Combination
Number analyzed (Participants) | 114 | 191
percentage of participants | 30.7 | 31.9
Statistical Analysis 1: Comparison: Biologic Monotherapy vs Biologic Combination; A two-sided Pearson's chi-squared test was used to assess the treatment difference in the participants who achieved DAS28 remission; Test type: Superiority or Other; p = 0.8222, Pearson's chi-squared; Treatment Difference = 1.2, 95% CI 2-sided [-9.5 to 12.0]

2. Secondary Outcome: Percentage of Participants Who Achieved DAS28-ESR Remission (DAS28-ESR <2.6) at 3 Months and at the Last Visit After Initiation of First-Line Biologic Treatment
Description: The DAS28 score is a measure of the participant's disease activity calculated using the TJC [28 joints], SJC [28 joints], participant's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the ESR for a total possible score of 0 to approximately 10. DAS28 = (0.56 * √ of TJC) + (0.28 * √ of SJC) + (0.70 * ln ESR in mm/h) + (0.014 * participant's global assessment of disease activity). DAS28 Remission is defined as a DAS28 score < 2.6.
Time Frame: Month 3 and the last visit (maximum 147.1 months for monotherapy and 189.1 months for combination therapy)
Population: Ten participants from all participants entered analysis set who could not be categorized as under biologic monotherapy or biologic combination therapy were excluded from analysis. Number of participants analyzed=participants with available data for DAS28-ESR. Here, 'n' signifies number of participants with available data for specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Biologic Monotherapy | Biologic Combination
Number analyzed (Participants) | 133 | 243
percentage of participants
  Month 3 (n=113,214) | 23.9 | 27.6
  Last visit (n=133,243) | 44.4 | 46.9
Statistical Analysis 1: Comparison: Biologic Monotherapy vs Biologic Combination; Comparison at Month 3. A two-sided Pearson's chi-squared test was used to assess the treatment difference in the participants who achieved DAS28 remission; Test type: Superiority or Other; p = 0.4727, Pearson's chi-squared; Treatment Difference = 3.7, 95% CI 2-sided [-6.2 to 13.6]
Statistical Analysis 2: Comparison: Biologic Monotherapy vs Biologic Combination; Comparison at last visit. A two-sided Pearson's chi-squared test was used to assess the treatment difference in the participants who achieved DAS28 remission; Test type: Superiority or Other; p = 0.6349, Pearson's chi-squared; Treatment Difference = 2.6, 95% CI 2-sided [-8.0 to 13.1]

3. Secondary Outcome: Percentage of Participants Who Achieved Low Disease Activity (LDA) (DAS28-ESR <3.2) at Months 3 and 6 and at the Last Visit After Initiation of First-Line Biologic Treatment.
Description: The DAS28 score is a measure of the participant's disease activity calculated using the TJC [28 joints], SJC [28 joints], participant's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the ESR for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. DAS28 Remission is defined as a DAS28 score <2.6. LDA was defined as a DAS28 score <3.2.
Time Frame: Months 3, 6 and last visit (maximum 147.1 months for monotherapy and 189.1 months for combination therapy)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Biologic Monotherapy | Biologic Combination
Number analyzed (Participants) | 133 | 243
percentage of participants
  Month 3 (n=113,214) | 42.5 | 41.6
  Month 6 (n=114,191) | 50.0 | 53.4
  Last visit (n=133,243) | 57.1 | 67.1
Statistical Analysis 1: Comparison: Biologic Monotherapy vs Biologic Combination; Comparison at Month 3. A two-sided Pearson's chi-squared test was used to assess the treatment difference in the participants who achieved LDA; Test type: Superiority or Other; p = 0.8769, Pearson's chi-squared; Slope = -0.9, 95% CI 2-sided [-12.1 to 10.4]
Statistical Analysis 2: Comparison: Biologic Monotherapy vs Biologic Combination; Comparison at Month 6. A two-sided Pearson's chi-squared test was used to assess the treatment difference in the participants who achieved LDA; Test type: Superiority or Other; p = 0.5649, Pearson's chi-squared; Treatment Difference = 3.4, 95% CI 2-sided [-8.2 to 15.0]
Statistical Analysis 3: Comparison: Biologic Monotherapy vs Biologic Combination; Comparison at the last visit. A two-sided Pearson's chi-squared test was used to assess the treatment difference in the participants who achieved LDA; Test type: Superiority or Other; p = 0.0556, Pearson's chi-squared; Treatment Difference = 9.9, 95% CI 2-sided [-0.3 to 20.2]

4. Secondary Outcome: Change From Baseline in DAS28 at Months 3, 6 and at The Last Visit After Initiation of First-Line Biologic Treatment
Description: The DAS28 score is a measure of the participant's disease activity calculated using the TJC [28 joints], SJC [28 joints], participant's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and either ESR or C Reactive Protein (CRP) for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. DAS28 Remission is defined as a DAS28 score <2.6.
Time Frame: Baseline, Month 3, 6 and last visit (maximum 147.1 months for monotherapy and 189.1 months for combination therapy)
Population: Ten participants from all participants entered analysis set who could not be categorized as under biologic monotherapy or biologic combination therapy were excluded from analysis. Number of participants analyzed=participants with post-baseline available data. Here, 'n' signifies number of participants with available data at specified category.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Biologic Monotherapy | Biologic Combination
Number analyzed (Participants) | 115 | 215
units on a scale
  Month 3 (n=103,198) | -2.74 (0.123) | -2.84 (0.089)
  Month 6 (n=105,180) | -3.00 (0.119) | -3.18 (0.089)
  Last visit (n=115,215) | -3.39 (0.124) | -3.54 (0.091)
Statistical Analysis 1: Comparison: Biologic Monotherapy vs Biologic Combination; Comparison at Month 3. Analysis used a mixed model with month, cohort, baseline DAS28 score; cohort-by-month and cohort-by-baseline DAS28 score as fixed effects. Within-participant repeated measurements were incorporated with an unstructured variance-covariance structure; Test type: Superiority or Other; p = 0.5195, Mixed Models Analysis; Treatment Difference = -0.10, 95% CI 2-sided [-0.40 to 0.20], Standard Error of Mean 0.152
Statistical Analysis 2: Comparison: Biologic Monotherapy vs Biologic Combination; Comparison at Month 6. Analysis used a mixed model with month, cohort, baseline DAS28 score; cohort-by-month and cohort-by-baseline DAS28 score as fixed effects. Within-participant repeated measurements were incorporated with an unstructured variance-covariance structure; Test type: Superiority or Other; p = 0.2420, Mixed Models Analysis; Treatment difference = -0.17, 95% CI 2-sided [-0.47 to 0.12], Standard Error of Mean 0.149
Statistical Analysis 3: Comparison: Biologic Monotherapy vs Biologic Combination; Comparison at the last visit. Analysis used a mixed model with month, cohort, baseline DAS28 score; cohort-by-month and cohort-by-baseline DAS28 score as fixed effects. Within-participant repeated measurements were incorporated with an unstructured variance-covariance structure; Test type: Superiority or Other; p = 0.3264, Mixed Models Analysis; Treatment difference = -0.15, 95% CI 2-sided [-0.45 to 0.15], Standard Error of Mean 0.154

5. Secondary Outcome: Percentage of Participants by Category of DAS28 Score and Timepoint
Description: The DAS28 score is a measure of the participant's disease activity calculated using the TJC [28 joints], SJC [28 joints], participant's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and either ESR or CRP for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. DAS28 Remission is defined as a DAS28 score <2.6.
Time Frame: Baseline, Month 3, 6 and last visit (maximum 147.1 months for monotherapy and 189.1 months for combination therapy)
Population: Ten participants from all participants entered analysis set who could not be categorized as under biologic monotherapy or biologic combination therapy were excluded from analysis. Number of participants analyzed=participants with available data for the endpoint. Here, 'n' signifies number of participants with available data for specifies category.
Measure: Number; unit: percentage of participants
Arm/Group | Biologic Monotherapy | Biologic Combination
Number analyzed (Participants) | 136 | 254
percentage of participants
  Baseline: <2.6 (n=117,219) | 2.6 | 0.5
  Baseline: ≥2.6 to ≤3.2 (n=117,219) | 0.9 | 0.5
  Baseline: >3.2 (n=117,219) | 96.6 | 99.1
  Baseline: >4 (n=117,219) | 95.7 | 98.2
  Month 3: <2.6 (n=117,222) | 24.1 | 27.9
  Month 3: ≥2.6 to ≤3.2 (n=117,222) | 19.8 | 17.6
  Month 3: >3.2 (n=117,222) | 56.0 | 54.5
  Month 3: >4 (n=117,222) | 37.1 | 32.9
  Month 6: <2.6 (n=117,200) | 29.9 | 30.5
  Month 6: ≥2.6 to ≤3.2 (n=117,200) | 23.1 | 24.5
  Month 6: >3.2 (n=117,200) | 47.0 | 45.0
  Month 6: >4 (n=117,200) | 29.9 | 22.5
  Last visit: <2.6 (n=136,254) | 44.1 | 46.9
  Last visit: ≥2.6 to ≤3.2 (n=136,254) | 18.4 | 23.2
  Last visit: >3.2 (n=136,254) | 37.5 | 29.9
  Last visit: >4 (n=136,254) | 20.6 | 15.4

6. Secondary Outcome: Duration of Treatment
Description: Drug retention was defined as the total duration of time in months the participant was on treatment (combination therapy or monotherapy). The duration was the time in months between the start date of biologic therapy to the date of most recent visit.
Time Frame: Baseline up to last visit (maximum 147.1 months for monotherapy and 189.1 months for combination therapy)
Population: Ten participants from all participants entered analysis set who could not be categorized as under biologic monotherapy or biologic combination therapy were excluded from analysis. Number of participants analyzed=participants with post-baseline available data for duration of treatment.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Biologic Monotherapy | Biologic Combination
Number analyzed (Participants) | 131 | 247
months | 57.30 (38.227) | 48.48 (34.619)
Statistical Analysis 1: Comparison: Biologic Monotherapy vs Biologic Combination; Analysis was performed using a general linear model with cohort as a factor; Test type: Superiority or Other; p = 0.0237, General Linear Model; Mean Difference (Final Values) = -8.81, 95% CI 2-sided [-16.44 to -1.18]

7. Secondary Outcome: Average Methotrexate Dose of Participants on Biological Combination Treatment
Time Frame: Baseline up to last visit (maximum 147.1 months for monotherapy and 189.1 months for combination therapy)
Population: Participants in biologic combination group from All Participants Entered Analysis Set. Number of participants analyzed=participants with available data for methotrexate dose.
Measure: Mean (Standard Deviation); unit: milligrams per week
Arm/Group | Biologic Combination
Number analyzed (Participants) | 178
milligrams per week | 17.12 (5.64)

8. Secondary Outcome: Change From Baseline in Total Number of Tender Joints at Months 3 and 6 and at the Last Visit After Initiation of First-Line Biologic Treatment.
Description: The 28 joints to be assessed for tenderness were shoulder, elbow, wrist, metacarpophalangeal (MCP) joints 1-5, proximal interphalangeal (PIP) joints 1-5, and knee on both sides of the body. The sum of tender joints ranged from 0 to 28 with 0 as best possible health status and 28 as worst health status.
Time Frame: Baseline, Month 3, 6 and last visit (maximum 147.1 months for monotherapy and 189.1 months for combination therapy)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Biologic Monotherapy | Biologic Combination
Number analyzed (Participants) | 129 | 245
tender joints
  Baseline (n=129,245) | 17.1 (6.98) | 16.3 (7.21)
  Change from baseline at Month 3 (n=106,203) | -12.5 (7.72) | -12.4 (6.95)
  Change from baseline at Month 6 (n=107,184) | -14.4 (6.93) | -13.4 (7.51)
  Change from baseline at Last visit (n=114,215) | -14.9 (8.18) | -14.3 (7.28)

9. Secondary Outcome: Change From Baseline in Total Number of Swollen Joints at Months 3 and 6 and at the Last Visit After Initiation of First-Line Biologic Treatment
Description: The 28 joints to be assessed for swelling were shoulder, elbow, wrist, MCP joints 1-5, PIP joints 1-5, and knee on both sides of the body. The sum of swollen joints, each, ranged from 0 to 28 with 0 as best possible health status and 28 as worst health status.
Time Frame: Baseline, Month 3, 6 and last visit (maximum 147.1 months for monotherapy and 189.1 months for combination therapy)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Biologic Monotherapy | Biologic Combination
Number analyzed (Participants) | 129 | 246
swollen joints
  Baseline (n=129,246) | 9.1 (5.27) | 10.0 (5.64)
  Change From Baseline at Month 3 (n=106,205) | -7.0 (5.05) | -7.2 (5.10)
  Change From Baseline at Month 6 (n=107,185) | -7.7 (5.24) | -8.3 (5.57)
  Change From Baseline at Last Visit (n=114,216) | -7.9 (5.73) | -8.8 (5.64)

ADVERSE EVENTS:
Time Frame: Baseline up to the last visit after initiation of first line biologic treatment (maximum 147.1 months for monotherapy and 189.1 months for combination therapy)
Description: Adverse events data were planned to be collected only for those participants who received rituximab or tocilizumab, as biologic therapy.
Groups:
- Biologic Monotherapy: Retrospective chart review of participants with RA who were being treated with first-line biologic drug therapy (only rituximab or tocilizumab) as monotherapy according to NICE guidelines.
- Biologic Combination: Retrospective chart review of participants with RA who were being treated with first-line biologic drug therapy (only rituximab or tocilizumab) plus MTX or biologic plus MTX plus any other classical DMARDs according to NICE guidelines.
Arm/Group | Biologic Monotherapy | Biologic Combination
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 0/7 | 2/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Biologic Monotherapy (N=7) | Biologic Combination (N=9)
Fatigue (General disorders) | 0 | 1
Influenza Like Illness (General disorders) | 0 | 1
Ear Pruritus (Ear and labyrinth disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Hot Flush (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.